CLINICAL TRIAL: NCT04972656
Title: Treatment With Ambrisentan in Patients With Borderline Pulmonary Arterial Hypertension: a Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Treatment With Ambrisentan in Patients With Borderline Pulmonary Arterial Hypertension
Acronym: TAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, HangZhang, Professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSC20210527
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambrisentan (Experimental): Monotherapy using ambrisentan will start at a dose of 5 mg (once daily) and will be up-titrated to 10 mg (once daily) after 4 weeks apart if patients are tolerable.
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Titration:
  Monotherapy using ambrisentan will be initialized at a beginning dose of 5 mg (once daily). Drug intake is scheduled at the morning. After 4 weeks monitoring, the dose of ambrisentan will be uptitrated to 10 mg once daily. Otherwise, if intolerability is indicated, a dose of 5 mg (once daily) will be maintained through the study duration.
  Maximum dose allowed: not to exceed 10 mg/day.
  Administration:
  Ambrisentan will be administered orally with or without food intake.
  Arms: Ambrisentan
Drug: Placebo — Placebo tablet (one to two tablets corresponding to one to two verum tablets).
  Administration:
  Placebo will be administrated orally with or without food intake in the morning.
  Arms: Placebo

SUMMARY:
An Investigator initiated trial (IIT) using a prospective, randomized, double-blind, parallel group, placebo-controlled, clinical study design.

DETAILED DESCRIPTION:
The treatment options and prognosis of patients with borderline pulmonary arterial hypertension (PAH) defined as mean pulmonary arterial pressure (mPAP) between 21-24 mm Hg measured by right heart catheterization (RHC) are understudied. The objective of this study is to determine the treatment effect of endothelin-receptor antagonist (Ambrisentan) for patients with borderline PAH when comparing with placebo. Accordingly, 420 patients with borderline PAH will be included in this prospective, randomized, double- blind, parallel group, placebo-controlled study. Repeat screening is required if last screening was performed > 30 days ago. Baseline medical history will be obtained and physical examination will be conducted before signed consent and randomization. Moreover, an electrocardiogram (ECG), laboratory testing, and transthoracic echocardiography (TTE) at supine will be carried out before randomization and during follow-up. Subjects have to meet all inclusion criteria and have no anyone of exclusion criteria. This study will comprise 3 stages: 1) screening period (0-30 days), 2) 1-year study period (365 ± 30 days), 3) extended follow-up duration 3 years ± 30 days. Repeat measurements of cardiac function, hemodynamic, exercise capacity, and clinical events will be scheduled at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be age ≥18 years;
* Subject has mPAP 21-24 mmHg, and PAWP<15mmHg.The underlying diseases that cause critical PAH belong to the first group, which is divided into: Idiopathic pulmonary hypertension, hereditary pulmonary hypertension, drugs and poisons associated with pulmonary hypertension, connective tissue diseases associated with pulmonary hypertension, HIV infection associated with pulmonary hypertension, portal hypertension associated with pulmonary hypertension, tumors associated with pulmonary hypertension, congenital heart disease associated with pulmonary hypertension.
* Subject (or legal guardian) understands the trial design and treatment procedures and provides written informal consent before any trial-specific tests or procedures are performed.

Exclusion Criteria:

* Pulmonary hypertension (PH) confirmed by right heart catheter (RHC) before enrolment, i.e. mPAP ≥25 mmHg at rest.
* Ongoing or a history of >2 weeks of continued use of therapies that are considered definitive PH treatment: endothelin receptor antagonists (ERA; e.g. bosentan, ambrisentan), phosphodiesterase type 5 inhibitors (PDE5; e.g. sildenafil, tadalafil, vardenafil), prostanoids (e.g. epoprostenol, treprostinil, iloprost, beraprost) and soluble guanylate cyclase stimulator (e.g. Riociguat). Intermittent use of PDE5 inhibitors for male erectile dysfunction is permitted.
* Known intolerance to ambrisentan or one of its excipients.
* Pulmonary vein occlusive disease
* Pulmonary capillary hemangiomatosis
* Surgical repair or interventional occlusion of congenital heart disease within 6 months prior to screening of this study
* Active connective tissue diseases
* Pulmonary hypertension due to left heart disease
* Pulmonary hypertension due to pulmonary disease and/or hypoxia
* Acute pulmonary embolism and/or chronic thromboembolism
* Clinically significant anemia, defined as hemoglobin concentration 75% below the normal lower limit.
* Renal insufficiency was defined as glomerular filtration rate [EGFR] <30 mL/min/1.73m2.
* Transaminase (ALT and/or AST) increased, exceeding the upper limit of normal value by 3 times.
* Arterial systolic blood pressure < 85 mmHg.
* Uncontrolled hypertension, defined as blood pressure >160/90 mmHg (resting state) and/or >220/120 mmHg (load state).
* Participate in any drug clinical trial within 4 weeks prior to screening in this study and/or plan to participate in another drug clinical trial during the study period.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of diagnostic PAH (mPAP ≥25 mmHg) | baseline, 1 year
  Determine whether mean pulmonary arterial pressure of patients with borderline - PAH (mPAP 21-24 mmHg) can be reduced by 3 mm Hg (absolute change baseline vs. 1 year; equals 15%) following treatment with ambrisentan 10 mg/die (initiated with 5 mg/die and elevated up to 10 mg/die) over 1 year (primary endpoint) compared to baseline and placebo.
Change of Pulmonary vascular resistance | baseline, 1 year
  Pulmonary vascular resistance by right heart catheterization

SECONDARY OUTCOMES:
Re-hospitalization due to clinical worsening | baseline, 3 years
  Re-hospitalization is defined as clinical manifestations of worsening PAH requiring re-hospitalization in order to add intravenous pharmacological agents (inotrope or vasodilator), mechanical intervention or ultrafiltration, hemofiltration, or dialysis.
All-cause mortality | baseline, 3 years
6-Minute-walking Test | baseline, 1 year
Right atrial pressure by right heart catheterization | baseline, 1 year
Cardiac output (CO) by right heart catheterization | baseline, 1 year
Cardiac index (CI) by right heart catheterization | baseline, 1 year
RA-area (right atrial area) by echocardiography | baseline, 1 year
RV-area (right ventricular area) by echocardiography | baseline, 1 year
Tei by echocardiography | baseline, 1 year
  Tei
TAPSE (tricuspid annular plane systolic excursion) by echocardiography | baseline, 1 year
sPAP (systolic pulmonary arterial pressure) by echocardiography | baseline, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China